CLINICAL TRIAL: NCT04888819
Title: A Multi-Center, Open-label, Randomized Trial to Evaluate the Efficacy and Safety Based on Timing of Administration of DWP14012 in Patients With Erosive Esophagitis
Brief Title: Treatment Effect According to Timing of Administration of DWP14012 40 mg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT_DWP14012001
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — fexuprazan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fed state group (Experimental): just after a meal
  Interventions: Drug: DWP14012
- fasted state group (Experimental): before a meal
  Interventions: Drug: DWP14012

INTERVENTIONS:
Drug: DWP14012 — DWP14012 40 mg, orally, once daily just after a meal up to 4 weeks
  Other Names: fed state
  Arms: fed state group
Drug: DWP14012 — DWP14012 40 mg, orally, once daily before a meal up to 4 weeks
  Other Names: fasted state
  Arms: fasted state group

SUMMARY:
The primary objective of this study is to establish noninferiority of efficacy of DWP14012 (40 mg once daily) based on Timing of Administration.

DETAILED DESCRIPTION:
Subjects will provide written informed consent for study participation and then undergo appropriate screening. Subjects who meet the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to either before meal group or after meal group. Subjects will be stratified into two groups according to Los Angeles classification grades (LA grades) A/B or C/D, as determined by upper gastrointestinal (GI) endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 19 and 75 years old based on the date of written agreement
* Those who have been diagnosed with erosive esophagitis of LA Grade A-D on the upper gastrointestinal endoscopy
* Those who experienced symptoms of heartburn or acid regurgitation within the last 7 days

Exclusion Criteria:

* Those who have undergone gastric acid suppression or gastric, esophageal surgery
* Those who with clinically significant liver, kidney, nervous system, respiratory, endocrine, hematologic, cardiovascular, urinary system disease

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
healing rate at week 4 | up to 4 weeks
  Cumulative healing rate of erosive esophagitis at week 4 by endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No